CLINICAL TRIAL: NCT02678130
Title: A Prospective Study of the InterFuse T(tm)
Brief Title: A Prospective Study of the InterFuse T(tm),
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vertebral Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-011
Record Dates: First submitted 2016-01-22; First posted 2016-02-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
Keywords: Intervertebral disc degeneration; Bone Disease; Musculoskeletal disease; Spinal disease
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Bone Diseases; Musculoskeletal Diseases; Spinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- InterFuse Group (Active Comparator): Patients are randomized based on last digit (odd) of social security number to be treated with an InterFuse T device
  Interventions: Device: InterFuse T
- Control Group: Standard of care TLIF (Active Comparator): treated with a standard of care TLIF (Transforaminal Lumbar Interbody Fusion) device (e.g. Stryker's AVS Unilif)
  Interventions: Device: Standard of Care TLIF (Stryker AVS Unilif)

INTERVENTIONS:
Device: InterFuse T — Transforaminal Lumbar Interbody fusion (TLIF)
  Arms: InterFuse Group
Device: Standard of Care TLIF (Stryker AVS Unilif) — Transforaminal Lumbar Interbody Fusion (TLIF)
  Arms: Control Group: Standard of care TLIF

SUMMARY:
The purpose of this post-approval study is to demonstrate that the InterFuse T modular lumbar interbody device is at least equal in safety and efficacy to other (standard of care) TLIF devices.

DETAILED DESCRIPTION:
The primary objective of this post-market study is to collect data to asses the long term outcome of the InterFuse T (tm) device in [patients undergoing interbody fusion.

The primary endpoints of the investigation will include assessment of the maintenance of disc height and fusion rates demonstrated by radiographic evidence based on plain radiographs. Fusion is defined as a bone bridging across the disc space at the level of the InterFuse T implant. Length of stay, implant migration, implant subsidence, re-operation rate and opioid use will be recorded. It is anticipated that outcomes with the InterFuse T Interbody Fusion Device will be comparable to or better than the historical published results for other non-modular TLIF devices and to the control device used concurrently in the study

ELIGIBILITY:
Inclusion Criteria:

* meets indications for an interbody fusion (determined by the study investigator)
* Has documented conservative (non-operative ) treatment for at least 3 months
* Has a VAS back pain of > or = 60mm
* Has an ODI > or = 40%
* at least 18 years of age and skeletally mature
* Willing and able to comply with study requirements
* Patient's condition is appropriate for surgery
* Agreed to participate in study

Exclusion Criteria:

* Has severe osteoporosis or osteopenia
* Grade 3 or higher Spondylolisthesis
* Diffuse multilevel neoplastic disease such that no adjacent normal segment exists for engagement or instrumentation
* Body Mass Index (BMI) > 40
* Patient has active infection
* Patient is pregnant or planning to become pregnant
* Patient is mentally ill or has history of drug abuse
* Patient has known allergy to Polyetheretherketone (PEEK), stainless steel or Tantalum
* Patient is currently enrolled in an investigational spine study
* Has rheumatoid arthritis, ankylosing spondylitis or other autoimmune disease
* patient bhas symptomatic fibrous arachnoiditis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
fusion rates | 12 months
  Assessment of the fusion rates as demonstrated by radiographic evidence.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | up to 12 months
  Visual Analog Scale pre-op compared to VAS score at 2-4 weeks, 6 months and at 1 year
Oswestry Disability Score (ODI) | 12 months
  Oswestry Low Back Pain Disability Questionaire
SF-36 | 12 months
  Rand 36-item Health Survey (version 1.0)
Maintenance of disk height | 12 months
  comparison of disk height pre-op versus at 12 months

OTHER OUTCOMES:
Length of hospital stay | up to 2-4 weeks
Opioid use | baseline, at 2-4 weeks, at 6 months and at 12 months
  usage of pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Kallhorn, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that data will be presented at scientific meetings and that a manuscript will be produced on the study